CLINICAL TRIAL: NCT06389071
Title: Safety and Efficacy of Ablative Fractional 2940 nm Laser Treatment for Lichen Sclerosus Lesion
Brief Title: Laser Treatment for Lichen Sclerosus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLS001
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lichen Sclerosus Lesion
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment + PRP Arm (Active Comparator)
  Interventions: Device: Fractional 2940 nm Laser
- Treatment only Arm (Active Comparator)
  Interventions: Device: Fractional 2940 nm Laser

INTERVENTIONS:
Device: Fractional 2940 nm Laser — Fractional 2940 nm Laser

SUMMARY:
Fractional ablative laser treatment for Lichen Sclerosus lesion

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years or older
* Biopsy-proven vulvar lichen sclerosus lesion
* Experiencing one or more of the following symptoms of LS:

  1. Dryness
  2. Itching
  3. Burning
  4. Bleeding
  5. Blistering
  6. Soreness
  7. Easily bruises
  8. Easily tears
  9. Ulcerated lesions
  10. Painful intercourse
* Negative urine pregnancy test if subject is of childbearing potential before enrollment
* Absence of vulvovaginal infection i.e. fungi, bacterial vaginosis, and STI
* Ability to understand and sign informed consent, questionnaires, and all investigation requirements
* Willing to consent to clinical photographs of the treatment area
* Willing to consent to ultrasound images of the treatment area
* Willing and able to logistically follow schedule of treatments and follow-up visits

Exclusion Criteria:

* Pregnancy, less than 3 months postpartum, or planning to become pregnant during the investigation to protect integrity of the data
* Is a nursing mother
* History of uncontrolled malignant disease
* Active urogenital infection or chronic infection (i.e., candida, herpes, herpes simplex, bacterial vaginosis, trichomoniasis, or other infection)
* Immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich syndrome)
* Subjects with genital skin disease, psoriasis due to risk of koeberizing
* Subjects on immunosuppressants: mycophenolate, retinoids, azathioprine, cyclosporin
* Known allergy or intolerance to local anesthesia
* Known history of connective tissue disease
* Known propensity for keloid formations
* Known medical condition that may affect wound healing
* Any reason that the investigator deems prohibits participation in the investigation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Histological clearance | 16 weeks
  Efficacy of the treatment is determined by histological changes measured at 16 weeks post final treatment

CONTACTS AND LOCATIONS:
Overall Officials: Josee Parent, MD, Principal Investigator — Clinique Medicale Uro-Gyneco de l'Abitibi
Locations (1):
- Clinique Medicale Uro-Gyneco de l'Abitibi, Val-d'Or, Quebec, Canada